CLINICAL TRIAL: NCT05768477
Title: Research of the Different Treatments for Chronic Pain Patients, Their Effectiveness and Associated Predictors, Offered at the Pain Center AZ Sint-Lucas Ghent.
Brief Title: Different Treatments in Chronic Pain Patients.
Acronym: EC_PC_AZSTL
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0090; 2021-39 (Registry Identifier: AZ Sint Lucas Hospital Ghent)
Record Dates: First submitted 2022-11-30; First posted 2023-03-14 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Nociplastic Pain
MeSH Terms: conditions — Chronic Pain; Nociplastic Pain | interventions — Referral and Consultation; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic pain patients: Chronic pain patients with a dominant nociceptive pain mechanism, a dominant neuropathic pain mechanism and a dominant nociplastic pain mechanism. They will receive different treatments: Consultations, Interventions (injections, denervations...), Baxter therapy and interdisciplinary treatment.
  Interventions: Other: Consultation; Procedure: Interventions; Drug: Baxter therapy; Behavioral: Interdisciplinary therapy

INTERVENTIONS:
Other: Consultation — Consultation with the pain specialist, which might entail prescription of medication of vitamins.
Procedure: Interventions — Facet injections, nerve denervations, infiltrations, Qutenza, Spinal Cord Stimulation, Transcutaneous Electrical Nerve Stimulation
Drug: Baxter therapy — Ketamine or Linisol baxter therapy
Behavioral: Interdisciplinary therapy — Interdisciplinary therapy provided by the physiotherapist, psychologist and occupational therapist.

SUMMARY:
The goal of this observational study is to compare different treatment options in a chronic pain population. The main questions it aims to answer are:

* What is the effectiveness of the different therapy options in the pain center of Sint-Lucas on outcomes related to pain and disability?
* What are predictive factors for the different therapy options in the pain center of Sint-Lucas? Which factors predict improvement in pain related outcomes?

Participant data will be gathered as part of their routine care. They can be advised to 4 different treatment options:

* Consultations with the pain specialist
* Interventions by the pain specialist (infiltrations, denervations)
* Baxter therapy
* Interdisciplinary treatment

Researchers will compare patients with different dominant pain mechanisms to see which treatment are most effective for which dominant pain mechanisms.

DETAILED DESCRIPTION:
The aim of the present study is to describe the natural flow of the chronic pain patients at the pain center AZ Sint-Lucas. Patients will be examined before starting the therapy, and receive standardized questionnaires at several fixed time points (before, during, and after their therapy trajectory). Information about the present dominant pain mechanism will be gathered during the examination. The questionnaires will gather demographic data, information about the present dominant pain mechanism, psychosocial factors, catastrophizing, fear and avoidance, illness perceptions, fatigue and information about therapy success. During the examination, typical signs of a dominant nociplastic pain mechanism will be gathered. By processing the data of the questionnaires and the examination, knowledge about (1) the amount of patients with a dominant nociplastic pain mechanism at intake, (2) the treatment trajectory for a specific diagnosis, and (3) the prediction of the therapy effect and prognosis will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Chronic pain patients
* Dutch speaking, or good understanding

Exclusion Criteria:

* Adults unable to give consent
* Adults who do not understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be patients attending the pain center of AZ Sint-Lucas in Ghent, a secondary care center for chronic pain patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain disability from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  Pain Disability Index, ranges from zero to 70, with a higher score indicating more pain-related disability
Change in Pain intensity from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  Numeric Rating Scale for pain intensity in the past week, ranges from zero to 100, with a higher score indicating a higher pain intensity
Change in Pain Frequency from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  Questions
Change in Functionality from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  Patient Specific Complaints questionnaire, using a Numeric Rating Scale, ranging from zero to 100, with a higher score indicating a higher amount of functional disability
Change in Quality of Life from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  EuroQol-5D questionnaire

SECONDARY OUTCOMES:
Change in Post exertional malaise from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  Questions based on the criteria for Chronic Fatigue Syndrome.
Change in Quality of Life from baseline until 18 months | 0 weeks, 4 weeks, 10 weeks, 6 months, 12 months, 18 months
  EuroQol - 5D, five questions about health range from one to three with a higher score indicating more difficulties. One question about perceived health ranges from zero to 100 with a higher score indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Principal Investigator — Department of Rehabilitation Sciences, Faculty of Health Sciences, Ghent University, Belgium
Locations (1):
- AZ St Lucas, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The personal data will be shared with the personal electronic patient file of AZ Sint-Lucas, of each patient.
  Sharing of data will be done upon reasonable request, and only for research purposes, after publication of the results. Data will be shared via a restricted data repository (FAIRsharing.org)
Time Frame: The data will not be transferred to a third country. The ethical committee of the pain center of AZ Sint-Lucas did not allow for data transfer upon reasonable request.
Access Criteria: The data will not be transferred to a third country.